CLINICAL TRIAL: NCT01549353
Title: Does Gum Chewing After Gynecologic Laparoscopy Stimulate Earlier Return of Bowel Motility?
Brief Title: Gum Chewing After Gynecologic Laparoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klinikum Klagenfurt am Wörthersee (Other)
Responsible Party: Principal Investigator, Husslein Heinrich, MD, Principal investigator, Klinikum Klagenfurt am Wörthersee
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: A 02/10
Record Dates: First submitted 2012-02-23; First posted 2012-03-09 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Postoperative Care
MeSH Terms: interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- chewing gum (Experimental)
  Interventions: Behavioral: gum chewing

INTERVENTIONS:
Behavioral: gum chewing

SUMMARY:
Gum chewing has been reported to stimulate bowel motility after open surgery, such as cesarean section and other abdominal surgeries. In general, after laparoscopic surgery problems with reduced bowel motility are not as common as after open surgery. In this study the investigators test the hypothesis that gum chewing is enhancing rapid return of bowel motility after gynecologic laparoscopic surgery. Further the investigators study patient satisfaction and potential side effects of postoperative gum chewing.

ELIGIBILITY:
Inclusion Criteria:

* all gynecologic laparoscopic surgery
* normal level of CA 125 postmenopausal

Exclusion Criteria:

* loose teeth
* chronic obstipation
* laparotomy
* operations longer then 3 h

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Time to return to active bowel movements | participants will be followed for the duration of hospital stay
  First active bowel movement is defined as time from operation until first passage of flatus. Time until first defecation will also be measured.

SECONDARY OUTCOMES:
patient satisfaction with postoperative gum chewing | participants will be followed for the duration of the hospital stay
  Satisfaction will be measured with a visual analog scale (1 participant would never chew gum postoperatively again - 10 participant would always like to chew gum postoperatively)
Number of participants with adverse events | participants will be followed for the duration of hospital stay
  All problems that are linked to postoperative gum chewing will be recorded (e.g. vomiting, aspiration,...)

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Klagenfurt am Woerthersee, Klagenfurt, Carinthia, Austria

REFERENCES:
- [Derived] Husslein H, Franz M, Gutschi M, Worda C, Polterauer S, Leipold H. Postoperative gum chewing after gynecologic laparoscopic surgery: a randomized controlled trial. Obstet Gynecol. 2013 Jul;122(1):85-90. doi: 10.1097/AOG.0b013e3182983e92. PMID 23743472